CLINICAL TRIAL: NCT00918268
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of Surface Antigen, Inactivated, Influenza Vaccine, Formulation 2009-2010, When Administered to Non-elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Surface Antigen, Inactivated, Influenza Vaccine Using the Strain Composition 2009/2010 Recommended in Northern Hemisphere in Non-elderly Adult and in Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71_10S; 2009-010598-19
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Influenza Disease
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (1):
- Influenza vaccine (Experimental)
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — One 0.5mL dose of Inactivated, Influenza Vaccine using the strain composition 2009/2010

SUMMARY:
Annual trial for registration influenza vaccine with the strain composition for season 2009/2010.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, mentally competent, willing and able to give written informed consent prior to study entry;
* able to comply with all the study requirements;
* in general good health as determined by:medical history, physical examination and- clinical judgment of the investigator Written informed consent must be obtained for all the subjects before enrollment into the study after the nature of the study has been explained.

Exclusion Criteria:

* They have any serious chronic or acute disease (in the judgment of the investigator) including but not limited to:

  1. Cancer, except for localized skin cancer;
  2. Advanced congestive heart failure
  3. Chronic obstructive pulmonary disease (COPD);
  4. Autoimmune disease (including rheumatoid arthritis);
  5. Acute or progressive hepatic disease;
  6. Acute or progressive renal disease;
  7. Severe neurological or psychiatric disorder
  8. Severe asthma
* They have history of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g., to ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin and neomycin sulphate);
* They have a known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting, for example, from:- receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study;receipt of immunostimulants,receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivates within the past 3 months and for the full length of the study and suspected or known HIV infection or HIV-related disease;
* They have a known or suspected history of drug or alcohol abuse;
* They have a bleeding diathesis or condition associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject;
* Female who are pregnant or nursing (breastfeeding) mothers or females of childbearing age do not plan to use acceptable birth control measures, for the duration of the study. Adequate contraception is defined as hormonal (e.g., oral, injection, transdermal patch, implant, cervical ring), barrier (e.g., condom or diaphragm), intrauterine device (IUD), or monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject's study entry;
* Within the past 12 months, they have:- received more than one injection of influenza vaccine
* Within the past 6 months, they have:-had laboratory confirmed influenza disease,- received influenza vaccine;
* Within the past 4 weeks they have received:-another vaccine;-any investigational agent;
* They have any acute or chronic infection requiring systemic antibiotic treatment or antiviral therapy within the last 7 days;
* They have experienced fever (i.e., axillary temperature≥ 38°C) within the last 3 days;
* They are taking part in another clinical study;
* They have any condition which, in the opinion of the investigator,might interfere with the evaluation of the study objectives;
* They are severely obese with Body Mass Index (BMI) > 35;
* Site personnel involved in the evaluation of safety and their immediate relatives are excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the antibody response to each influenza vaccine antigen, as measured by Single Radial Hemolysis (SRH) at 21 days post-immunization in non-elderly adult and elderly subjects | 21(-1/+5) days
Evaluation of safety of a single intramuscular injection of influenza vaccine in non elderly adult and elderly subjects | 21(-1/+5) days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- Italy (3):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G. D'Annunzio, Via dei Vestini, Chieti
  - Ufficio Igiene e Sanità Pubblica di Lanciano, ASL Lanciano - Vasto, sede legale Via S. Spaventa, 37 ----- Satellite sites: (a) Distretto Sanitario di Base, Via Don Minzoni, Lanciano (CH) and (b) Distretto Sanitario di Base, Via Polidoro, Fossacesia (CH)), Lanciano
  - Pianiga Distretto n. 2 - Area Sud - Azienda ULSS 13 Mirano-Via Nazionale 48, Pianiga